CLINICAL TRIAL: NCT02295267
Title: Molecular Analysis of IgE Antibodies in Walnut Allergic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Paul Ehrlich Institute Langen (Unknown); Hospital Clinic of Barcelona (Other); St. Marien Hospital Bonn (Unknown); Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2012-0519
Record Dates: First submitted 2014-11-11; First posted 2014-11-20 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Food Allergy
Keywords: Food allergy; Walnut; Components; Allergens
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- walnut allergy provocation (Experimental): inclusion of walnut allergic patients, food provocation with walnut
  Interventions: Other: walnut allergy provocation

INTERVENTIONS:
Other: walnut allergy provocation — double blind placebo controlled food challenge

SUMMARY:
Accurate diagnosis of food allergy depends on the identification of the causative allergenic molecule(s). The proposed study intends to investigate and compare the pattern of IgE antibody sensitisation in walnut allergic subjects from three different regions of Europe (south (SEU) and central/north (C/NEU), to evaluate the diagnostic utility of a panel of novel allergen reagents.

DETAILED DESCRIPTION:
Accurate diagnosis of food allergy depends on the identification of the causative allergenic molecule(s). Thus, full characterization of the major allergens of walnut and their clinical importance is an important undertaking.

The proposed study intends to investigate and compare the pattern of IgE antibody sensitisation in walnut allergic subjects from three different regions of Europe (south (SEU) and central/north (C/NEU), to evaluate the diagnostic utility of a panel of novel allergen reagents.

With a view towards improved in vitro diagnostic methods, we intend to evaluate the diagnostic potential of recombinant walnut allergens in patients with walnut allergy confirmed by a positive provocation or supported by a convincing history of anaphylactic reaction(s) to walnut in the past, patients with pollinosis but no symptoms of walnut allergy and non-atopic control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Group A: positive case history of allergic reaction(s) to walnut
* Group B: positive case history of allergy to birch, grass or olive pollen and no case history of allergic reaction(s) to walnut
* Group C: no case history of atopic disease

Exclusion Criteria:

* Known pregnancy
* Breast-feeding of infant
* Treatment with the following drugs (or shortest interval between last treatment and food challenge or SPT):
* corticosteroids (2 weeks): applied systemically, to the nose or locally on the skin test area.
* antihistamines (3 days) except hydroxyzine (10 days)
* betablocker agents (1 day)
* angiotensin converting enzyme inhibitors (2 days)
* Any major organic or infectious disease

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-12; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
numbers of patients with walnut allergy | December 2012 to November 2017, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ballmer-Weber, PI, Principal Investigator — Allergy Unit, Department of Dermatology, University Zürich
Locations (1):
- Allergy Unit, Department of Dermatology, University Hospital, Zurich, Switzerland